CLINICAL TRIAL: NCT02136836
Title: Investigation of the Proportion of Human Epidermal Growth Factor Receptor 2 Protein Overexpression of Gastric Adenocarcinoma and Prognostic Effect of HER2, and Analysis of Practice Pattern of Herceptin Use in Stage IV Gastric Cancer
Acronym: HER2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jae Yong Cho, Chief of division of medical oncology, Gangnam Severance Hospital, Yonsei University
Other Study IDs: GSCH-STO13-01; Roche (Other: Roche)
Record Dates: First submitted 2014-05-08; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Stomach Neoplasms
Keywords: Genes, erbB-2; Prognosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- gastric adenocarcinoma

SUMMARY:
The objective of this study is to investigate the proportion of HER2 overexpression in gastric cancer patients group, to evaluate the relation of HER2 overexpression with prognosis, and to analyze the proportion of herceptin applied to patients in clinical field. Furthermore, the investigators are going to reevaluate the clinical benefit of Herceptin for survival prolongation compared to chemotherapy only.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma
2. Patients were diagnosed during 2006-2013
3. HER2 expression status was evaluated in primary gastric cancer or metastatic lesion.

Exclusion Criteria:

* Patients with second primary cancer within 5 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: gastric cancer patients in Gangnam Severance Hospital
Sampling Method: Non-Probability Sample
Enrollment: 860 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of HER2 overexpression in gastric cancer patients | 8 years

SECONDARY OUTCOMES:
Gastric cancer specific survival according to HER2 expression in each stage | 5 years

OTHER OUTCOMES:
The practice pattern of Herceptin use in stage IV gastric cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Cho, M.D.,Ph.D., Principal Investigator — Gangnam Severance Hospital, Yonsei University
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea